CLINICAL TRIAL: NCT05830500
Title: A Real World Study of Anlotinib for Patients With Advanced Medullary Thyroid Carcinoma
Brief Title: Study of Anlotinib in Patients With Advanced Medullary Thyroid Carcinoma
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ALOT-MTC-1
Record Dates: First submitted 2023-04-14; First posted 2023-04-26 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-04

CONDITIONS: Medullary Thyroid Cancer
MeSH Terms: conditions — Carcinoma, Medullary

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anlotinib capsules (Experimental): Anlotinib: 12 mg once daily for 2 weeks, followed by a discontinuance of 1 week (21-daya as a cycle)
  Interventions: Drug: Anlotinib Hydrochloride Capsule
- Observation (No Intervention): Observational group: prospectively and retrospectively collect data for patients who did not receive anlotinib hydrochloride capsules or similar small-molecule antivascular inhibitors (including Rearranged during transfection (RET) inhibitors, etc.).

INTERVENTIONS:
Drug: Anlotinib Hydrochloride Capsule — Anlotinib hydrochloride is a muti-target tyrosine kinase inhibitor that inhibits both tumor angiogenesis and tumor cell proliferation simultaneously.
  Arms: Anlotinib capsules

SUMMARY:
This is a real world study aiming to observe the efficacy and safety of Anlotinib capsules in patients with advanced medullary thyroid carcinoma, and to summarize the treatment experience in a broad population of patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients voluntarily joined the study, signed the informed consent, and had good compliance;
* Patients ≥18 years of age (at the time of signing the informed consent); Eastern Cooperative Oncology Group Performance Status (ECOG-PS) score: 0-2; Expected survival of more than 3 months;
* Patients were pathologically confirmed as inoperable locally advanced or metastatic medullary thyroid carcinoma (MTC), possessing imaging or clinical evidence of disease progression within the first 14 months of enrollment;
* Having at least one measurable lesion (assessed by Response Evaluation Criteria In Solid Tumors (RECIST) 1.1);
* Major organ functions meet the following criteria within 7 days prior to the treatment:

  1. Blood routine examination shall meet the following standards (no transfusion within 14 days) :

     1. Hemoglobin (Hb) ≥85g/L;
     2. Absolute Neutrophil Count (ANC) ≥1.5×109/L;
     3. Platelet (PLT) ≥80×109/L；
  2. Biochemical examination shall meet the following standards:

     1. Total bilirubin (TBIL) ≤1.5 times the upper limit of normal (ULN);
     2. Alanine transferase (ALT) and Aspartate transferase (AST) ≤2.5×ULN; If accompanied by liver metastasis, ALT and AST ≤5×ULN；
     3. Serum creatinine (Cr) ≤1.5×ULN or Creatinine clearance rate (CCr) ≥60ml/min；
* Female patients of reproductive age should agree that birth control (such as intrauterine device, birth control pills, or condoms) must be used during the study period until six months after completion; Having a negative serum pregnancy test within 7 days prior to study enrollment, and must be non-lactating; Male patients should agree to use contraception during the study period until six months after the end of the study.

Exclusion Criteria:

* Complicated diseases and history:

  1. Patients currently have or had other malignancies within 3 years. Patients with the following two conditions can be included in the group: Continuous 5-year disease-free survival (DFS) was achieved for other malignancies treated with a single operation. Cured cervical carcinoma in situ, non-melanoma skin cancer, and superficial bladder tumors [Ta (non-invasive tumor), Tis (carcinoma in situ) and T1 (the tumor infiltrates the basal membrane)];
  2. Major surgical treatment, open biopsy, or significant traumatic injury were received within 28 days before the beginning of the treatment;
  3. Subjects with any severe and/or uncontrolled disease, including:

     1. Having ≥ grade 2 myocardial ischemia or myocardial infarction or arrhythmia (including QTc ≥450ms (male), QTc ≥470ms (female) and ≥ grade 2 congestive heart failure (classified by New York heart association, NYHA));
     2. Active or uncontrolled severe infection (≥ Common Terminology Criteria for Adverse Events (CTC AE) 2 grade of infection);
     3. Renal failure requiring hemodialysis or peritoneal dialysis;
* Patients with concomitant diseases that, in the investigator's judgment, may seriously endanger patients' safety or may interfere with the completion of the study, or are deemed unsuitable for inclusion for other reasons.
* Patients who have previously used anlotinib hydrochloride capsules or similar Vascular Endothelial Growth Factor- Tyrosine Kinase Inhibitor (VEGFR-TKI) small molecule drugs, such as vandetanib, cabozantinib, lenvatinib, sunitinib, sorafenib, etc.;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2023-06-19 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | Baseline up to 3 years.
  The proportion of subjects who achieves a best overall response of complete response (CR) or partial response (PR).
Progression-free Survival (PFS) | Baseline up to 3 years.
  From the first dose of investigational drug to the date of disease progression or death, whichever occurs first.

SECONDARY OUTCOMES:
Disease-control Rate (DCR) | Baseline up to 3 years.
  The proportion of subjects response of CR, PR, or stable disease (SD) (subjects achieving SD will be included in the DCR if they maintain SD for ≥4 weeks).
Duration of Response (DOR) | Baseline up to 3 years.
  From the date that CR or PR are first occurred to the date of disease progression or death, whichever occurs first.
Overall Survival (OS) | Baseline up to death event, up to 3 years.
  From randomization to the time of death from any cause.
Adverse event rate | Baseline up to 3 years.
  The occurrence of all adverse events (AEs), serious adverse events (SAEs) and treatment-related adverse events (TEAEs).

CONTACTS AND LOCATIONS:
Locations (19):
- China (19):
  - Anhui Provincial Cancer Hospital, Hefei, Anhui
  - Beijing Tongren Hospital Affiliated to Capital Medical University, Beijing, Beijing Municipality
  - Gansu Cancer Hospital, Lanzhou, Gansu
  - Guangxi Zhuang Autonomous Region Cancer Hospital (Affiliated Cancer Hospital of Guangxi Medical University), Nanning, Guangxi
  - The First Affiliated Hospital of Hebei North University, Shijiazhuang, Hebei
  - Tianjin Cancer Hospital, Tianjin, Hebei
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - Nanjing Drum Tower Hospital The Affiliated Hospital of Nanjing University, Nanjing, Jiangsu
  - Jiangsu North People's Hospital, Yangzhou, Jiangsu
  - Liaoning Cancer Hospital and Institute, Shenyang, Liaoning
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi’an, Shanxi
  - Shanxi Provincial Tumor Hospital, Xi’an, Shanxi
  - Tianjin People's Hospital, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang